CLINICAL TRIAL: NCT00229008
Title: A Phase 3 Randomized Double-Blind Study Of Ceftobiprole Medocaril Versus Linezolid Plus Ceftazidime In The Treatment Of Nosocomial Pneumonia
Brief Title: Ceftobiprole in Hospital Acquired Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR005140; BAP00248
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Pneumonia
Keywords: Ceftobiprole medocaril; Nosocomial Pneumonia; Ventilator-Associated Pneumonia; Cephalosporins; Methicillin-Resistant Staphylococcus Aureus
MeSH Terms: conditions — Pneumonia; Healthcare-Associated Pneumonia; Pneumonia, Ventilator-Associated | interventions — ceftobiprole; Linezolid; Ceftazidime

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 001 (Experimental): ceftobiprole plus placebo ceftobiprole 500 mg every 8 hours as a 120 minute intravenous infusion and placebo administered every 12 hours as a 60-minute intravenous infusion for 7 to 14 days
  Interventions: Drug: ceftobiprole plus placebo
- 002 (Active Comparator): linezolid plus ceftazidime linezolid 600 mg every 12 hours as a 60-minute intravenous infusion plus ceftazidime 2 g every 8 hours as a 120-minute intravenous infusion for 7 to 14 days
  Interventions: Drug: linezolid plus ceftazidime

INTERVENTIONS:
Drug: ceftobiprole plus placebo — ceftobiprole 500 mg every 8 hours as a 120 minute intravenous infusion and placebo administered every 12 hours as a 60-minute intravenous infusion for 7 to 14 days
  Arms: 001
Drug: linezolid plus ceftazidime — linezolid 600 mg every 12 hours as a 60-minute intravenous infusion plus ceftazidime 2 g every 8 hours as a 120-minute intravenous infusion for 7 to 14 days
  Arms: 002

SUMMARY:
The purpose of this study is to compare the clinical cure rate of ceftobiprole medocaril (the water-soluble prodrug [form] of ceftobiprole) referred to as ceftobiprole versus a comparator in the treatment of patients with nosocomial pneumonia.

DETAILED DESCRIPTION:
Ceftobiprole medocaril (the water-soluble prodrug [form] of ceftobiprole) referred to as ceftobiprole is a cephalosporin antibiotic with anti-MRSA (Methicillin-Resistant Staphylococcus Aureus) activity. Ceftobiprole is not yet approved for the treatment of nosocomial (hospital-acquired) pneumonia. This is a randomized, double-blind, multicenter study of ceftobiprole versus a comparator (linezolid plus ceftazidime) to assess the effectiveness and safety of ceftobiprole in patients with nosocomial pneumonia. The patients will be randomized to ceftobiprole plus placebo or the comparator. The primary endpoint is the clinical cure rate of ceftobiprole at the test-of-cure visit. The patients will receive either ceftobiprole plus placebo or the comparator for 7 to 14 days (unless extended at discretion of medical monitor). Patient safety will be monitored throughout the study. In December 2006, this study (BAP00248) and another similar study (BAP00307, see NCT00210964) were amended (changed) to create 1 study (BAP00248/307).Therefore, the results reported for this study will be combined with the results reported for study BAP00248 Patients will receive either ceftobiprole plus placebo or a comparator by intravenous infusion for 7 to 14 days (unless extended at discretion of medical monitor).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from nosocomial pneumonia or ventilator-associated pneumonia
* Female patients must be postmenopausal for at least 1 year, surgically sterile, or practicing an effective method of birth control, before entry and throughout the study, and have a negative serum or urine pregnancy test at the screening

Exclusion Criteria:

* Known or suspected hypersensitivity to any related antibiotic medications
* Any known or suspected condition or concurrent treatment that would be contraindicated by the prescribing information
* Treatment with any investigational drug within 30 days before enrollment
* Prior enrollment to this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-11; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Clinical cure rate (the ratio of the number of clinically cured patients to the total number of patients in the population) | 7 to 14 days after the end of therapy (EOT)

SECONDARY OUTCOMES:
Microbiological eradication rate | At the TOC visit defined as 7-14 days after the EOT
Clinical cure rate | At the late follow-up (LFU) visit defined as 28 to 35 days after the EOT
Microbiological eradication rates | At the LFU visit defined as 28 to 35 days after the EOT
Pneumonia-specific mortality rates | Within 30 days after the randomization

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Huang H, Gao L, Engelhardt M, Saulay M, Hamed K. A post hoc analysis of two Phase III trials showing the efficacy and tolerability of ceftobiprole in East Asian patients. Future Microbiol. 2021 Jul;16:783-796. doi: 10.2217/fmb-2021-0121. Epub 2021 Jun 22. PMID 34155899
- [Derived] Welte T, Scheeren TW, Overcash JS, Saulay M, Engelhardt M, Hamed K. Efficacy and safety of ceftobiprole in patients aged 65 years or older: a post hoc analysis of three Phase III studies. Future Microbiol. 2021 May;16:543-555. doi: 10.2217/fmb-2021-0042. Epub 2021 May 7. PMID 33960817
- [Derived] Scheeren TWL, Welte T, Saulay M, Engelhardt M, Santerre-Henriksen A, Hamed K. Early improvement in severely ill patients with pneumonia treated with ceftobiprole: a retrospective analysis of two major trials. BMC Infect Dis. 2019 Feb 26;19(1):195. doi: 10.1186/s12879-019-3820-y. PMID 30808293
- [Derived] Awad SS, Rodriguez AH, Chuang YC, Marjanek Z, Pareigis AJ, Reis G, Scheeren TW, Sanchez AS, Zhou X, Saulay M, Engelhardt M. A phase 3 randomized double-blind comparison of ceftobiprole medocaril versus ceftazidime plus linezolid for the treatment of hospital-acquired pneumonia. Clin Infect Dis. 2014 Jul 1;59(1):51-61. doi: 10.1093/cid/ciu219. Epub 2014 Apr 9. PMID 24723282
- See also: Ceftobiprole in Hospital Acquired Pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=635&filename=CR005032_CR005140_CSR.pdf